CLINICAL TRIAL: NCT03316547
Title: Supporting and Enhancing NICU Sensory Experiences to Optimize Developmental Outcomes in Preterm Infants
Brief Title: Supporting and Enhancing NICU Sensory Experiences (SENSE)
Acronym: SENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201601057
Record Dates: First submitted 2017-08-15; First posted 2017-10-20 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Premature Birth of Newborn
Keywords: preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: SENSE program-treatment; standard-of-care-control
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Parents were asked to participate in a study investigating 2 different approaches to sensory exposures in the NICU. The approach (SENSE or standard of care) were described after enrollment, based on which group they were randomized to. The evaluator was blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group received standard hospital care.
- Intervention (Experimental): Parents in the sensory-based intervention group were educated to provide daily sensory-based interventions across the length of hospitalization as outlined in the manualized intervention (the SENSE Program). A sensory support team completed the doses of sensory exposures when parents were unable.
  Interventions: Other: SENSE Program

INTERVENTIONS:
Other: SENSE Program — Specific amounts of auditory, tactile, vestibular, kinesthetic, and visual exposure conducted daily through hospitalization. This includes specifically timed and set amounts of reading/talking/singing, cycled lighting, skin-to-skin (kangaroo) care or gentle human touch, rocking, and therapeutic exercises [passive range of motion (PROM), gentle stretching]. The intervention plan is intended to be implemented by parents when available, and by surrogates when the parents are unable to be present in the hospital. Specific amounts and timing of interventions will be tailored to the current medical status and age of each infant.
  Other Names: Sensory-Based Intervention
  Arms: Intervention

SUMMARY:
Seventy preterm infants born less than or equal to 32 weeks gestation were put into either the sensory-based intervention (experiment) group or traditional care (control) group. Consecutive admissions at St. Louis Children's Hospital (SLCH) who were hospitalized in a private NICU room were recruited. The parents of infants in the sensory-based intervention group were educated and supported by trained therapists to give different positive sensory experiences to their infants while hospitalized. The traditional care group received normal, standard care while hospitalized. For both care groups, infant neurobehavior, sensory processing, and parent mental health were measured at term age prior to hospital discharge. Child development, sensory processing, and parent mental health were measured again at age one year (corrected). Differences between the two groups were explored.

DETAILED DESCRIPTION:
Approximately 12%, or 500,000 infants, are born preterm each year in the United States alone. Although survival rates of preterm infants have increased with advances in medical care, the risk of developmental delay and disability has remained constant. Very preterm infants (<32 weeks gestation) necessitate care in the neonatal intensive care unit (NICU) for an average of three months after birth, which is a significant period of time coinciding with a critical window of brain development. While medical factors, such as brain injury, can heighten the risk of adverse neurodevelopmental outcome, the NICU environment may also have deleterious effects on early brain structure and function.

The Influence of Early Environment: Maternal deprivation and isolation from positive sensory experiences are prominent features of orphan studies. Consequences of language and human deprivation include emotional disturbances, delayed cognitive and language skills, and abnormalities evident on magnetic resonance imaging (MRI). Although the preterm infant differs from a child who has been institutionalized or deprived of caregiving attention after full term birth, there are similarities, such as the altered temporal lobe structures, and the pattern of developmental impairments. There is growing evidence supporting the importance of parents in the NICU. Low frequency visits between parents and their hospitalized preterm infants have been associated with suboptimal outcomes, like child abuse and abandonment and adverse emotional functioning. NICU's in Sweden have been successful with engaging parents in care from admission to discharge and have reported shorter hospitalizations. There is also a growing body of evidence supporting positive sensory exposures for preterm infants, including maternal voice recordings, massage, skin-to-skin holding, and vestibular and kinesthetic interventions. In addition, my team has made important research findings pointing to the potential need for developmentally-appropriate sensory exposures in the NICU.

Outcomes Associated with Preterm Birth: While advances in medical technologies have improved the rates of survival among preterm infants, the risk of long-term morbidities remains high, with 50-70% of very preterm infants exhibiting developmental problems. In addition to motor problems, language and communication problems are common in former preterm infants when studied at school age, and recent evidence suggests that language deficits persist through childhood. Language difficulties have also been shown to affect a broad range of factors important for social prowess and academic achievement. In addition, preterm infants have a heightened risk of attachment disorders and other social-emotional problems.

Outcomes Associated with Parenting a Preterm Infant: Many negative psychological sequelae are associated with parenting a preterm infant, including depression, anxiety, and post-traumatic stress. Such negative parental mental health outcomes proceed to influence the parent-child relationship, leading to a parent's inability to recognize infant cues as well as increased negativity and intrusiveness. Negative maternal-child interactions continue into the first several months of life if stress remains high. Forming such a foundation may then lead to negative child outcomes associated with social-emotional development, including attachment insecurity, and mental health issues.

Sensory Stimuli and Current Practice in the NICU: High-risk infants who receive care in the NICU are exposed to significant stressors that include painful procedures, disruption of normal sensory experiences, and stress related to parent-infant separation. In addition to the loss of parental nurturing, there is growing concern that stress during a period of extensive brain development may result in permanent and deleterious developmental outcomes.

Developmental care, which includes sensory minimization, has been the predominant model of care in the NICU since the 1980s, because the bright and noisy environment, which exceeds sensory standards set by the American Academy of Pediatrics, is understood to adversely affect growth and development of the preterm infant. In support of developmental care principles, NICU staff makes efforts to reduce modifiable stimuli to the high-risk infant in the NICU. However, there is emerging research on the positive effects of sensory stimulation for preterm infants in the NICU.

Positive sensory exposures in the NICU are critical, as they can have life-long implications on learning, memory, emotions, and developmental progression. In an environment where stimuli are primarily negative, it is especially important to define and implement positive sensory exposures in the NICU. Further, it is well understood that multi-dimensional sensory exposures are present in utero in the final months and weeks of pregnancy, but the preterm infant misses potentially important, timed exposures that may be absent or altered in the NICU environment. Positive forms of sensory exposure during periods of infant readiness may be important to facilitate appropriate neural pathways and enable positive experiences.

Results from a rigorous systematic review, benchmarking, and expert opinion were used to develop a clinical practice guideline for sensory-based interventions for hospitalized, very preterm infants using the Appraisal of Guidelines for Research and Evaluation II instrument. The manualized intervention (from the integrative review and development of the implementation plan) includes evidenced-based interventions that can be conducted by parents with their preterm infants across postmenstrual age while hospitalized. The sensory-based intervention includes the provision of specific amounts of auditory, tactile, vestibular, kinesthetic, olfactory, and visual exposure to be conducted daily through hospitalization. The intervention plan is intended to be implemented by parents (when available) and by surrogates when the parents are unable to be present in the hospital. Surveys, focus groups of a multidisciplinary team of health care professionals and parents of preterm infants in the NICU, and a pilot/feasibility study were conducted to assess acceptability, appropriateness and feasibility of the sensory-based intervention plan. The investigators enrolled 30 very preterm infants within the first week of life and implemented the sensory-based program. Logging sheets were placed at the infant's bedside to document the execution of sensory-based interventions, who conducted the intervention (parent, member of research team or other caregiver), and infant responses and consequences of the intervention. Physiological (such as heart rate and oxygen saturation fluctuations), state (levels of arousal) and behavioral (such as crying, changes in motoric tone) responses were recorded by caregivers during interventions on the bedside logs. Negative sequelae of the intervention resulted in stopping the intervention and modifying the criteria for sensory-based interventions accordingly. A licensed therapist provided guidance as to when infants can and cannot tolerate sensory exposures. From clinical documentation and bedside logging, implementation factors were assessed. Adaptations to the sensory-based program were made until it was deemed appropriate by the investigative team. This occurred after the model for an enhanced sensory environment could be documented 75% of the time on at least 3 consecutive participants.

The aim of this randomized clinical trial was to assess the effect of a sensory-based intervention in the NICU on outcomes of preterm infants and their families.

After obtaining informed consent, 70 preterm infants were randomized to 2 levels of sensory exposure: the sensory-based intervention or traditional care group. The parents of infants in the sensory-based intervention group were educated and supported to conduct sensory interventions with their infants using the systematized protocol. The traditional care group had therapists and nurses provide and educate parents about sensory exposures as standard of care. For both care groups, infant neurobehavior, sensory processing, mother-infant interaction, and parent mental health were assessed at term age prior to hospital discharge. Child development, sensory processing, and parent mental health were measured again at age one year corrected using standardized measures. Differences between groups were explored.

ELIGIBILITY:
Inclusion Criteria:

Preterm Infants:

* A prospective cohort very preterm infants (VPT) born less than or equal to 32 weeks gestation at the St. Louis Children's Hospital in St. Louis, Missouri.
* Infant is less than or equal to 7 days old when approached about the study.

Parents:

-Parents (including emancipated minors age 12-17) of very preterm infants (VPT) born less than or equal to 32 weeks gestation at the St. Louis Children's Hospital in St. Louis, Missouri.

Exclusion Criteria:

Preterm Infants:

* Known or suspected congenital anomaly, congenital infection (e.g., syphilis, HIV, TORCH), or known prenatal brain lesions (e.g., cysts or infarctions)
* Infants that are wards of the state, or become wards of the state after enrolling in the study. Any data collected beginning at the time the state obtains custody onward will not be used in the research study.
* Infants who are in the open ward area/bed spaces of the SLCH NICU (due to the significant variation in sensory exposure among those infants, and also to provide consistency during the hospital's impending transition to strictly private rooms in the very near future).

Parents:

-Parents with limited or no understanding of the English Language

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta G Pineda, PhD, OTR/L, Principal Investigator — Washington University School of Medicine; University of Southern California
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Volpe, J., Neurology of the Newborn 2008, Saunders: Philadelphia.
- [Background] Seay B, Harlow HF. Maternal separation in the rhesus monkey. J Nerv Ment Dis. 1965 Jun;140(6):434-41. doi: 10.1097/00005053-196506000-00006. No abstract available. PMID 4953280
- [Background] Tottenham N, Hare TA, Quinn BT, McCarry TW, Nurse M, Gilhooly T, Millner A, Galvan A, Davidson MC, Eigsti IM, Thomas KM, Freed PJ, Booma ES, Gunnar MR, Altemus M, Aronson J, Casey BJ. Prolonged institutional rearing is associated with atypically large amygdala volume and difficulties in emotion regulation. Dev Sci. 2010 Jan 1;13(1):46-61. doi: 10.1111/j.1467-7687.2009.00852.x. PMID 20121862
- [Background] Tottenham N, Sheridan MA. A review of adversity, the amygdala and the hippocampus: a consideration of developmental timing. Front Hum Neurosci. 2010 Jan 8;3:68. doi: 10.3389/neuro.09.068.2009. eCollection 2009. PMID 20161700
- [Background] BRODBECK AJ, IRWIN OC. The speech behaviour of infants without families. Child Dev. 1946 Sep;17(3):145-56. No abstract available. PMID 20285787
- [Background] Govindan RM, Behen ME, Helder E, Makki MI, Chugani HT. Altered water diffusivity in cortical association tracts in children with early deprivation identified with Tract-Based Spatial Statistics (TBSS). Cereb Cortex. 2010 Mar;20(3):561-9. doi: 10.1093/cercor/bhp122. Epub 2009 Jun 22. PMID 19546156
- [Background] Aeby A, Van Bogaert P, David P, Baleriaux D, Vermeylen D, Metens T, De Tiege X. Nonlinear microstructural changes in the right superior temporal sulcus and lateral occipitotemporal gyrus between 35 and 43 weeks in the preterm brain. Neuroimage. 2012 Oct 15;63(1):104-10. doi: 10.1016/j.neuroimage.2012.06.013. Epub 2012 Jun 17. PMID 22713672
- [Background] Barre N, Morgan A, Doyle LW, Anderson PJ. Language abilities in children who were very preterm and/or very low birth weight: a meta-analysis. J Pediatr. 2011 May;158(5):766-774.e1. doi: 10.1016/j.jpeds.2010.10.032. Epub 2010 Dec 10. PMID 21146182
- [Background] Reynolds LC, Duncan MM, Smith GC, Mathur A, Neil J, Inder T, Pineda RG. Parental presence and holding in the neonatal intensive care unit and associations with early neurobehavior. J Perinatol. 2013 Aug;33(8):636-41. doi: 10.1038/jp.2013.4. Epub 2013 Feb 14. PMID 23412640
- [Background] Fanaroff AA, Kennell JH, Klaus MH. Follow-up of low birth weight infants--the predictive value of maternal visiting patterns. Pediatrics. 1972 Feb;49(2):287-90. No abstract available. PMID 5059535
- [Background] Latva R, Lehtonen L, Salmelin RK, Tamminen T. Visiting less than every day: a marker for later behavioral problems in Finnish preterm infants. Arch Pediatr Adolesc Med. 2004 Dec;158(12):1153-7. doi: 10.1001/archpedi.158.12.1153. PMID 15583100
- [Background] Ortenstrand A, Westrup B, Brostrom EB, Sarman I, Akerstrom S, Brune T, Lindberg L, Waldenstrom U. The Stockholm Neonatal Family Centered Care Study: effects on length of stay and infant morbidity. Pediatrics. 2010 Feb;125(2):e278-85. doi: 10.1542/peds.2009-1511. Epub 2010 Jan 25. PMID 20100748
- [Background] Krueger C, Parker L, Chiu SH, Theriaque D. Maternal voice and short-term outcomes in preterm infants. Dev Psychobiol. 2010 Mar;52(2):205-12. doi: 10.1002/dev.20426. PMID 20112262
- [Background] Diego MA, Field T, Hernandez-Reif M. Preterm infant weight gain is increased by massage therapy and exercise via different underlying mechanisms. Early Hum Dev. 2014 Mar;90(3):137-40. doi: 10.1016/j.earlhumdev.2014.01.009. Epub 2014 Jan 27. PMID 24480603
- [Background] Hernandez-Reif M, Diego M, Field T. Preterm infants show reduced stress behaviors and activity after 5 days of massage therapy. Infant Behav Dev. 2007 Dec;30(4):557-61. doi: 10.1016/j.infbeh.2007.04.002. Epub 2007 Jun 4. PMID 17548111
- [Background] Mendes EW, Procianoy RS. Massage therapy reduces hospital stay and occurrence of late-onset sepsis in very preterm neonates. J Perinatol. 2008 Dec;28(12):815-20. doi: 10.1038/jp.2008.108. Epub 2008 Jul 17. PMID 18633421
- [Background] Feldman R, Rosenthal Z, Eidelman AI. Maternal-preterm skin-to-skin contact enhances child physiologic organization and cognitive control across the first 10 years of life. Biol Psychiatry. 2014 Jan 1;75(1):56-64. doi: 10.1016/j.biopsych.2013.08.012. Epub 2013 Oct 4. PMID 24094511
- [Background] Scher MS, Ludington-Hoe S, Kaffashi F, Johnson MW, Holditch-Davis D, Loparo KA. Neurophysiologic assessment of brain maturation after an 8-week trial of skin-to-skin contact on preterm infants. Clin Neurophysiol. 2009 Oct;120(10):1812-8. doi: 10.1016/j.clinph.2009.08.004. Epub 2009 Sep 17. PMID 19766056
- [Background] White-Traut RC, Nelson MN, Silvestri JM, Vasan U, Littau S, Meleedy-Rey P, Gu G, Patel M. Effect of auditory, tactile, visual, and vestibular intervention on length of stay, alertness, and feeding progression in preterm infants. Dev Med Child Neurol. 2002 Feb;44(2):91-7. doi: 10.1017/s0012162201001736. PMID 11848115
- [Background] Vignochi CM, Silveira RC, Miura E, Canani LH, Procianoy RS. Physical therapy reduces bone resorption and increases bone formation in preterm infants. Am J Perinatol. 2012 Sep;29(8):573-8. doi: 10.1055/s-0032-1310520. Epub 2012 Jul 6. PMID 22773291
- [Background] Maguire CM, Walther FJ, van Zwieten PH, Le Cessie S, Wit JM, Veen S. Follow-up outcomes at 1 and 2 years of infants born less than 32 weeks after Newborn Individualized Developmental Care and Assessment Program. Pediatrics. 2009 Apr;123(4):1081-7. doi: 10.1542/peds.2008-1950. PMID 19336365
- [Background] Reproductive Health, Preterm Birth. March 23, 2012; Available from: http://www.cdc.gov/reproductivehealth/maternalinfanthealth/PretermBirth.htm.
- [Background] Williams J, Lee KJ, Anderson PJ. Prevalence of motor-skill impairment in preterm children who do not develop cerebral palsy: a systematic review. Dev Med Child Neurol. 2010 Mar;52(3):232-7. doi: 10.1111/j.1469-8749.2009.03544.x. Epub 2010 Feb 4. PMID 20002114
- [Background] Botting, N., Z. Simkin, and G. Conti-Ramsden, Associated reading skills in children with a history of Specific Language Impairment (SLI). Read Writ, 2006. 19: p. 77-98.
- [Background] Durkin K, Conti-Ramsden G. Language, social behavior, and the quality of friendships in adolescents with and without a history of specific language impairment. Child Dev. 2007 Sep-Oct;78(5):1441-57. doi: 10.1111/j.1467-8624.2007.01076.x. PMID 17883441
- [Background] Mulder H, Pitchford NJ, Hagger MS, Marlow N. Development of executive function and attention in preterm children: a systematic review. Dev Neuropsychol. 2009;34(4):393-421. doi: 10.1080/87565640902964524. PMID 20183707
- [Background] Pedespan L. [Attachment and prematurity]. Gynecol Obstet Fertil. 2004 Sep;32(9):716-20. doi: 10.1016/j.gyobfe.2004.06.016. French. PMID 15380751
- [Background] Quesada AA, Tristao RM, Pratesi R, Wolf OT. Hyper-responsiveness to acute stress, emotional problems and poorer memory in former preterm children. Stress. 2014 Sep;17(5):389-99. doi: 10.3109/10253890.2014.949667. PMID 25089937
- [Background] Miles MS, Holditch-Davis D, Schwartz TA, Scher M. Depressive symptoms in mothers of prematurely born infants. J Dev Behav Pediatr. 2007 Feb;28(1):36-44. doi: 10.1097/01.DBP.0000257517.52459.7a. PMID 17353730
- [Background] Zelkowitz P, Na S, Wang T, Bardin C, Papageorgiou A. Early maternal anxiety predicts cognitive and behavioural outcomes of VLBW children at 24 months corrected age. Acta Paediatr. 2011 May;100(5):700-4. doi: 10.1111/j.1651-2227.2010.02128.x. Epub 2011 Jan 11. PMID 21214883
- [Background] Holditch-Davis D, Bartlett TR, Blickman AL, Miles MS. Posttraumatic stress symptoms in mothers of premature infants. J Obstet Gynecol Neonatal Nurs. 2003 Mar-Apr;32(2):161-71. doi: 10.1177/0884217503252035. PMID 12685667
- [Background] O'Hara MW, McCabe JE. Postpartum depression: current status and future directions. Annu Rev Clin Psychol. 2013;9:379-407. doi: 10.1146/annurev-clinpsy-050212-185612. Epub 2013 Feb 1. PMID 23394227
- [Background] Spinelli M, Poehlmann J, Bolt D. Predictors of parenting stress trajectories in premature infant-mother dyads. J Fam Psychol. 2013 Dec;27(6):873-83. doi: 10.1037/a0034652. Epub 2013 Nov 4. PMID 24188086
- [Background] Shah PE, Clements M, Poehlmann J. Maternal resolution of grief after preterm birth: implications for infant attachment security. Pediatrics. 2011 Feb;127(2):284-92. doi: 10.1542/peds.2010-1080. Epub 2011 Jan 17. PMID 21242223
- [Background] Woodward LJ, Bora S, Clark CA, Montgomery-Honger A, Pritchard VE, Spencer C, Austin NC. Very preterm birth: maternal experiences of the neonatal intensive care environment. J Perinatol. 2014 Jul;34(7):555-61. doi: 10.1038/jp.2014.43. Epub 2014 Mar 20. PMID 24651730
- [Background] Gray RF, Indurkhya A, McCormick MC. Prevalence, stability, and predictors of clinically significant behavior problems in low birth weight children at 3, 5, and 8 years of age. Pediatrics. 2004 Sep;114(3):736-43. doi: 10.1542/peds.2003-1150-L. PMID 15342847
- [Background] Nomura Y, Wickramaratne PJ, Warner V, Mufson L, Weissman MM. Family discord, parental depression, and psychopathology in offspring: ten-year follow-up. J Am Acad Child Adolesc Psychiatry. 2002 Apr;41(4):402-9. doi: 10.1097/00004583-200204000-00012. PMID 11931596
- [Background] Smith GC, Gutovich J, Smyser C, Pineda R, Newnham C, Tjoeng TH, Vavasseur C, Wallendorf M, Neil J, Inder T. Neonatal intensive care unit stress is associated with brain development in preterm infants. Ann Neurol. 2011 Oct;70(4):541-9. doi: 10.1002/ana.22545. Epub 2011 Oct 4. PMID 21976396
- [Background] Douret, L., M. Robin, and M. Le Normandy, The history of care of premature infants: from neonate intensive care to special care baby unit. Early Child Dev Care, 1994. 182: p. 21-29.
- [Background] Noise: a hazard for the fetus and newborn. American Academy of Pediatrics. Committee on Environmental Health. Pediatrics. 1997 Oct;100(4):724-7. No abstract available. PMID 9836852
- [Background] Brandon DH, Holditch-Davis D, Belyea M. Preterm infants born at less than 31 weeks' gestation have improved growth in cycled light compared with continuous near darkness. J Pediatr. 2002 Feb;140(2):192-9. doi: 10.1067/mpd.2002.121932. PMID 11865270
- [Background] Field T. Alleviating stress in newborn infants in the intensive care unit. Clin Perinatol. 1990 Mar;17(1):1-9. PMID 2180616
- [Background] Graven SN, Bowen FW Jr, Brooten D, Eaton A, Graven MN, Hack M, Hall LA, Hansen N, Hurt H, Kavalhuna R, et al. The high-risk infant environment. Part 1. The role of the neonatal intensive care unit in the outcome of high-risk infants. J Perinatol. 1992 Jun;12(2):164-72. No abstract available. PMID 1522437
- [Background] Byers JF. Components of developmental care and the evidence for their use in the NICU. MCN Am J Matern Child Nurs. 2003 May-Jun;28(3):174-80; quiz 181-2. doi: 10.1097/00005721-200305000-00007. PMID 12771696
- [Background] Lasky RE, Williams AL. Noise and light exposures for extremely low birth weight newborns during their stay in the neonatal intensive care unit. Pediatrics. 2009 Feb;123(2):540-6. doi: 10.1542/peds.2007-3418. PMID 19171620
- [Background] Lickliter R. The integrated development of sensory organization. Clin Perinatol. 2011 Dec;38(4):591-603. doi: 10.1016/j.clp.2011.08.007. Epub 2011 Oct 13. PMID 22107892
- [Background] Hepper PG, Shahidullah BS. Development of fetal hearing. Arch Dis Child Fetal Neonatal Ed. 1994 Sep;71(2):F81-7. doi: 10.1136/fn.71.2.f81. PMID 7979483
- [Background] Pineda RG, Stransky KE, Rogers C, Duncan MH, Smith GC, Neil J, Inder T. The single-patient room in the NICU: maternal and family effects. J Perinatol. 2012 Jul;32(7):545-51. doi: 10.1038/jp.2011.144. Epub 2011 Oct 27. PMID 22031044
- [Background] Pineda, R., Neil, J., Dierker, D., Smyser, C., Kidokora, H., Reynolds, L., Walker, S., Rogers, C., Mathur, A., VanEssen, D., Inder, T., The Impact of Different Neonatal Intensive Care Environments on Brain Development and Function in Preterm Infants, 2012, Washington University School of Medicine.
- [Background] Caskey, M., Tucker, R., Vohr. Language environment in a single familly room NICU. in Pediatric Academic Societies. 2012. Boston, MA.
- [Background] Liu WF. Comparing sound measurements in the single-family room with open-unit design neonatal intensive care unit: the impact of equipment noise. J Perinatol. 2012 May;32(5):368-73. doi: 10.1038/jp.2011.103. Epub 2011 Aug 18. PMID 21852773
- [Background] Brouwers MC, Kho ME, Browman GP, Burgers JS, Cluzeau F, Feder G, Fervers B, Graham ID, Grimshaw J, Hanna SE, Littlejohns P, Makarski J, Zitzelsberger L; AGREE Next Steps Consortium. AGREE II: advancing guideline development, reporting and evaluation in health care. J Clin Epidemiol. 2010 Dec;63(12):1308-11. doi: 10.1016/j.jclinepi.2010.07.001. Epub 2010 Jul 24. No abstract available. PMID 20656455
- [Background] Pineda JA, Leonard JR, Mazotas IG, Noetzel M, Limbrick DD, Keller MS, Gill J, Doctor A. Effect of implementation of a paediatric neurocritical care programme on outcomes after severe traumatic brain injury: a retrospective cohort study. Lancet Neurol. 2013 Jan;12(1):45-52. doi: 10.1016/S1474-4422(12)70269-7. Epub 2012 Nov 28. PMID 23200264
- [Background] Proctor EK, Powell BJ, Baumann AA, Hamilton AM, Santens RL. Writing implementation research grant proposals: ten key ingredients. Implement Sci. 2012 Oct 12;7:96. doi: 10.1186/1748-5908-7-96. PMID 23062065
- [Background] Proctor E. Implementation science and child maltreatment: methodological advances. Child Maltreat. 2012 Feb;17(1):107-12. doi: 10.1177/1077559512437034. Epub 2012 Feb 15. No abstract available. PMID 22337867
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Proctor EK, Landsverk J, Aarons G, Chambers D, Glisson C, Mittman B. Implementation research in mental health services: an emerging science with conceptual, methodological, and training challenges. Adm Policy Ment Health. 2009 Jan;36(1):24-34. doi: 10.1007/s10488-008-0197-4. Epub 2008 Dec 23. PMID 19104929
- [Background] Proctor EK, Rosen A. From Knowledge Production to Implementation: Research Challenges and Imperatives. Res Soc Work Pract. 2008 Jul 1;18(4):285-291. doi: 10.1177/1049731507302263. PMID 24089591
- [Background] Khlif MS, Colditz PB, Boashash B. Effective implementation of time-frequency matched filter with adapted pre and postprocessing for data-dependent detection of newborn seizures. Med Eng Phys. 2013 Dec;35(12):1762-9. doi: 10.1016/j.medengphy.2013.07.005. Epub 2013 Aug 21. PMID 23972955
- [Background] Lobb R, Colditz GA. Implementation science and its application to population health. Annu Rev Public Health. 2013;34:235-51. doi: 10.1146/annurev-publhealth-031912-114444. Epub 2013 Jan 7. PMID 23297655
- [Background] Wolin KY, Colditz GA, Proctor EK. Maximizing benefits for effective cancer survivorship programming: defining a dissemination and implementation plan. Oncologist. 2011;16(8):1189-96. doi: 10.1634/theoncologist.2011-0054. Epub 2011 Jul 17. PMID 21765196
- [Background] Speilberger, C., State-Trait Anxiety Inventory for Adults. 2005-2008, Menlo Park, CA: Mind Garden.
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Endler, N., Coping Inventory for Stressful Situations (CISS): Manual. 1990, Toronto: Multi-Health Systems.
- [Background] Abidin, R.R., Parenting stress index professional manual. 3 ed. 1995, Odessa, FL: Psychological Assessment Resources, Inc.
- [Background] Tronick E, Lester BM. Grandchild of the NBAS: the NICU network neurobehavioral scale (NNNS): a review of the research using the NNNS. J Child Adolesc Psychiatr Nurs. 2013 Aug;26(3):193-203. doi: 10.1111/jcap.12042. PMID 23909942
- [Background] Dunn, W., Infant/Toddler Sensory Profile 2. 2014, San Antonio: Pearson Education, Inc.
- [Background] Squires, J., et al., Ages and Stages Questionnaires - 3. 2009, Baltimore, MD: Paul H. Brookes Publishing Co.
- [Background] Beck, A.T., R.A. Steer, and G.K. Brown, Manual for the beck depression inventory-II. 1996, San Antonio, TX: Psychological Corporation.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Snaith, R.P. and A.S. Zigmond, The hospital anxiety and depression scale manual. 1994, Windsor, Ontario: NFER-Nelson.
- [Background] Yu YT, Hsieh WS, Hsu CH, Chen LC, Lee WT, Chiu NC, Wu YC, Jeng SF. A psychometric study of the Bayley Scales of Infant and Toddler Development - 3rd Edition for term and preterm Taiwanese infants. Res Dev Disabil. 2013 Nov;34(11):3875-83. doi: 10.1016/j.ridd.2013.07.006. Epub 2013 Sep 9. PMID 24029804
- [Result] Pineda RG, Tjoeng TH, Vavasseur C, Kidokoro H, Neil JJ, Inder T. Patterns of altered neurobehavior in preterm infants within the neonatal intensive care unit. J Pediatr. 2013 Mar;162(3):470-476.e1. doi: 10.1016/j.jpeds.2012.08.011. Epub 2012 Oct 1. PMID 23036482
- [Result] Howe TH, Sheu CF, Wang TN, Hsu YW. Parenting stress in families with very low birth weight preterm infants in early infancy. Res Dev Disabil. 2014 Jul;35(7):1748-56. doi: 10.1016/j.ridd.2014.02.015. Epub 2014 Mar 19. PMID 24656293
- [Result] Singer LT, Fulton S, Kirchner HL, Eisengart S, Lewis B, Short E, Min MO, Satayathum S, Kercsmar C, Baley JE. Longitudinal predictors of maternal stress and coping after very low-birth-weight birth. Arch Pediatr Adolesc Med. 2010 Jun;164(6):518-24. doi: 10.1001/archpediatrics.2010.81. PMID 20530301
- [Result] Wraight CL, McCoy J, Meadow W. Beyond stress: describing the experiences of families during neonatal intensive care. Acta Paediatr. 2015 Oct;104(10):1012-7. doi: 10.1111/apa.13071. Epub 2015 Jun 26. PMID 26058331
- [Result] Bouet KM, Claudio N, Ramirez V, Garcia-Fragoso L. Loss of parental role as a cause of stress in the neonatal intensive care unit. Bol Asoc Med P R. 2012 Jan-Mar;104(1):8-11. PMID 22788072
- [Result] Heinemann AB, Hellstrom-Westas L, Hedberg Nyqvist K. Factors affecting parents' presence with their extremely preterm infants in a neonatal intensive care room. Acta Paediatr. 2013 Jul;102(7):695-702. doi: 10.1111/apa.12267. Epub 2013 May 8. PMID 23590800
- [Result] Anderson P, Doyle LW; Victorian Infant Collaborative Study Group. Neurobehavioral outcomes of school-age children born extremely low birth weight or very preterm in the 1990s. JAMA. 2003 Jun 25;289(24):3264-72. doi: 10.1001/jama.289.24.3264. PMID 12824207
- [Result] Anderson PJ, Doyle LW. Cognitive and educational deficits in children born extremely preterm. Semin Perinatol. 2008 Feb;32(1):51-8. doi: 10.1053/j.semperi.2007.12.009. PMID 18249240
- [Result] Holsti L, Grunau RV, Whitfield MF. Developmental coordination disorder in extremely low birth weight children at nine years. J Dev Behav Pediatr. 2002 Feb;23(1):9-15. doi: 10.1097/00004703-200202000-00002. PMID 11889346
- [Result] Goyen TA, Lui K, Woods R. Visual-motor, visual-perceptual, and fine motor outcomes in very-low-birthweight children at 5 years. Dev Med Child Neurol. 1998 Feb;40(2):76-81. doi: 10.1111/j.1469-8749.1998.tb15365.x. PMID 9489494
- [Result] Pineda RG, Neil J, Dierker D, Smyser CD, Wallendorf M, Kidokoro H, Reynolds LC, Walker S, Rogers C, Mathur AM, Van Essen DC, Inder T. Alterations in brain structure and neurodevelopmental outcome in preterm infants hospitalized in different neonatal intensive care unit environments. J Pediatr. 2014 Jan;164(1):52-60.e2. doi: 10.1016/j.jpeds.2013.08.047. Epub 2013 Oct 17. PMID 24139564
- [Result] Bystron I, Blakemore C, Rakic P. Development of the human cerebral cortex: Boulder Committee revisited. Nat Rev Neurosci. 2008 Feb;9(2):110-22. doi: 10.1038/nrn2252. PMID 18209730
- [Result] Burns CM, Rutherford MA, Boardman JP, Cowan FM. Patterns of cerebral injury and neurodevelopmental outcomes after symptomatic neonatal hypoglycemia. Pediatrics. 2008 Jul;122(1):65-74. doi: 10.1542/peds.2007-2822. PMID 18595988
- [Result] Berument SK, Sonmez D, Eyupoglu H. Supporting language and cognitive development of infants and young children living in children's homes in Turkey. Child Care Health Dev. 2012 Sep;38(5):743-52. doi: 10.1111/j.1365-2214.2011.01314.x. Epub 2011 Sep 27. PMID 21951265
- [Result] Daunhauer LA, Coster WJ, Tickle-Degnen L, Cermak SA. Effects of caregiver-child interactions on play occupations among young children institutionalized in Eastern Europe. Am J Occup Ther. 2007 Jul-Aug;61(4):429-40. doi: 10.5014/ajot.61.4.429. PMID 17685176
- [Result] Daunhauer LA, Coster WJ, Tickle-Degnen L, Cermak SA. Play and cognition among young children reared in an institution. Phys Occup Ther Pediatr. 2010 May;30(2):83-97. doi: 10.3109/01942630903543682. PMID 20367513
- [Result] Ellis BH, Fisher PA, Zaharie S. Predictors of disruptive behavior, developmental delays, anxiety, and affective symptomatology among institutionally reared romanian children. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1283-92. doi: 10.1097/01.chi.0000136562.24085.160. PMID 15381896

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 39 | 31
Completed | 21 | 18
Not Completed | 18 | 13
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Transfer to another hospital | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 39 | 31 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 31 | 70
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: EGA at birth (weeks)] | 29.5 (2.5) | 29.7 (2.6) | 29.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 19 | 47
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 18 | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 31 | 70

OUTCOME MEASURES:

1. Primary Outcome: Ages and Stages Questionnaire (ASQ) - Communication at 1 Year
Description: Parents completed the parent-report measure of child development, the Ages and Stages Questionnaire (ASQ), at 1 year corrected age. The ASQ The Communication subscore is the primary variable of interest, which looks at the child's language and communication skills at time of assessment. Higher scores on the ASQ Communication subsection indicate more positive outcomes. A child can score a minimum of 0 points and a maximum of 60 points on the Communication subscale.
Time Frame: One year corrected age
Population: As noted in Participant Flow module, overall number of participants analyzed reflects participants who completed testing at 1 year follow-up (decrease in participants due to death, transfer, and loss to follow-up).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 21 | 18
score on a scale | 38.6 (18.1) | 48.6 (10.3)

2. Primary Outcome: Neonatal Intensive Care Unit (NICU) Network Neurobehavioral Scale (NNNS) Excitability Score at Term Equivalent Age
Description: Infants were assessed using the NICU Network Neurobehavioral Scale (NNNS) by a blinded evaluator. The Excitability subscore, which measures state-related level of arousal over the course of the whole examination, is the primary variable of interest, and ranges from 1-8. An average response falls in the moderate, midpoint range (4-5), and describes an infant who could be brought to respond to stimuli in spite of a high degree of upset or excitement, but then can return to moderate state. Thus, a midpoint range score (4-5) would indicate a better outcome on the Excitability sub scale, whereas a lower (<4) or higher (>5) score would indicate a worse outcome.
Time Frame: At term equivalent age (35-41 weeks PMA)
Population: Overall number of participants analyzed reflects number of participants assessed at term equivalent age (some were lost at this time point for this assessment due to death or transfer to a different hospital).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: The control group received standard hospital care.
  N = 39
- Intervention: Parents in the sensory-based intervention group were educated to provide daily sensory-based interventions across the length of hospitalization as outlined in the manualized intervention (the SENSE Program). A sensory support team completed the doses of sensory exposures when parents were unable.
  SENSE Program: Specific amounts of auditory, tactile, vestibular, kinesthetic, and visual exposure conducted daily through hospitalization. This includes specifically timed and set amounts of reading/talking/singing, cycled lighting, skin-to-skin (kangaroo) care or gentle human touch, rocking, and therapeutic exercises [passive range of motion (PROM), gentle stretching]. The intervention plan is intended to be implemented by parents when available, and by surrogates when the parents are unable to be present in the hospital. Specific amounts and timing of interventions will be tailored to the current medical status and age of each infant.
  N = 31
Arm/Group | Control | Intervention
Number analyzed (Participants) | 28 | 24
score on a scale | 4.4 (2.7) | 4.1 (2.2)

3. Secondary Outcome: Language Environmental Acquisition Device (LENA)
Description: Audio recordings of a single 16 hour period to capture language and sound exposure occurred at 34 weeks using the Language Environmental Acquisition Device (LENA). The LENA device is a digital language processor that captures environmental sound for up to 16 hours and quantifies: % of the recording with meaningful word exposure, % of the recording with electronic noise, % of the recording with noise, % of the recording with silence, and % of the recording with distant word exposure.
Time Frame: Single 16 hour period to capture language and sound exposure will occur at 34 weeks to assess treatment fidelity/differentiation.
Population: Overall number of participants analyzed reflects number of participants assessed at 34 weeks (some were lost at this time point for this assessment due to death or transfer to a different hospital or inability to complete recording due to technological or administrative issues).
Measure: Mean (Standard Deviation); unit: percentage of 16h recording
Arm/Group | Control | Intervention
Number analyzed (Participants) | 17 | 12
percentage of 16h recording
  % Meaningful words | 2.4 (1.5) | 3.9 (3.0)
  % Distant words | 2.6 (2.6) | 3.7 (2.6)
  % TV or electronic sounds | 14.8 (14.0) | 14.3 (17.4)
  % Noise | 12.5 (9.7) | 10.2 (9.1)
  % Silence | 67.7 (17.8) | 68.0 (18.5)

4. Secondary Outcome: Sensory Exposures Provided During Hospitalization
Description: During each day of hospitalization (from day of consent, often within 1 week of birth, to day of discharge, often near term-equivalent age; an average of about 2 months), parents, health care professionals and the sensory support team documented the type and amount of tactile and auditory exposures conducted. The proportion of the SENSE program doses, whether parents conducted the majority of the sensory exposures and whether the doses were met were defined after hospital discharge was complete.
Time Frame: Sensory exposures were documented every day of hospitalization (from birth to term-equivalent age; an average of about 2 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 28 | 24
Participants
  # of infants who received > 75% of recommended doses of sensory interventions | 14 | 24
  # of infants who received 100% of recommended doses of sensory interventions | 8 | 15
  Parent provided > 50% of interventions received | 12 | 12

5. Secondary Outcome: Dubowitz/Hammersmith Neonatal Neurological Evaluation
Description: At the NICU bedside, infant neurobehavior was assessed by a blinded evaluator using the Dubowitz/Hammersmith Neonatal Neurological Evaluation (HNNE). The HNNE is an assessment of neonatal neurological status. The total score is used as an outcome variable and ranges from 0-78. A higher score indicates a better outcome, whereas a lower score indicates a worse outcome.
Time Frame: At term equivalent age (between 35-41 weeks post menstrual age), just prior to discharge from the hospital.
Population: The number of participants analyzed reflects the number of infants who underwent HNNE assessment at 35-41 weeks post menstrual age; some infants were not assessed at this time point due to death or transfer to a different hospital prior to NICU discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 28 | 24
score on a scale | 22.8 (4.0) | 20.6 (3.4)

6. Secondary Outcome: General Movement Assessment (GMA)
Description: A video recording was conducted to enable scoring of general movements and infant neurological/motor status using the General Movements Assessment. However, video quality was deemed insufficient for analysis.
Time Frame: At term equivalent age (between 35-41 weeks post menstrual age), just prior to discharge from the hospital.
Population: Video quality was insufficient for appropriate scoring and thus not analyzed.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Discharge Questionnaire
Description: Prior to discharge from the hospital, the infant's mother completed a questionnaire. Measures included the Sensory Profile-2 (SP-2), the State Trait Anxiety Inventory (STAI), the Edinburgh Postnatal Depression Scale (EPDS), the Parent Stress Index (PSI), The Parental Stress Scale: NICU (PSS), the Maternal Confidence Questionnaire, and the Infant Care Questionnaire (ICQ). The SP-2 assesses infant sensory processing skills with summary scores for tactile, auditory, visual, movement, oral, and general processing. The STAI measures maternal anxiety separated into state-related and trait-related anxiety. The PSI includes subscales to measure defensive responding, parental distress, parent-child dysfunctional interaction, & difficult child behaviors. The ICQ measures maternal connection, emotionality, and responsiveness. Possible score ranges and directions of scores listed with each variable below.
Time Frame: Just prior to discharge from the hospital (between 35-41 weeks post menstrual age).
Population: Questionnaires were included if complete; number of participants analyzed reflects number of completed questionnaires. Reasons for questionnaire incompletion were: infant death, transfer prior to discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 28 | 24
score on a scale
  Sensory Profile - Touch (range 3-15) - higher = possible dysfunction | 4.3 (1.8) | 4.8 (2.1)
  Sensory Profile - Auditory (range 4-20) higher = possible dysfunction | 9.2 (3.7) | 8.1 (3.4)
  Sensory Profile - Visual (range 4-20)higher = possible dysfunction | 6.7 (4.0) | 5.6 (2.8)
  Sensory Profile - Movement (range 4-20) higher = possible dysfunction | 8.0 (2.0) | 7.9 (2.4)
  Sensory Profile - Oral (range 2-10) higher = possible dysfunction | 4.6 (1.9) | 4.2 (1.7)
  Sensory Profile - General (range 8-40) higher = possible dysfunction | 14.1 (5.7) | 14.9 (5.6)
  PSI- Defensive Responding (range 7-35) Higher = more dysfunction | 13.3 (5.4) | 13.0 (6.1)
  PSI - Parental Distress (range 12-60) Higher = more dysfunction | 22.7 (7.7) | 22.6 (10.0)
  PSI - Parent-Child Dysfunctional Interaction (range 12-60) Higher = more dysfunction | 19.6 (5.4) | 18.7 (7.5)
  PSI - Difficult Child (range 12-60) Higher = more dysfunction | 18.2 (5.2) | 17.4 (5.7)
  Edinburgh Postnatal Depression Scale (range 0-30) Higher = more likelihood of depression | 9.0 (4.7) | 8.5 (5.5)
  Parental Stressor Scale - NICU (range 0-5), Higher = more stress | 3.1 (1.2) | 2.5 (1.0)
  STAI - State Anxiety (range 20-80) Higher = more anxiety | 38.5 (11.9) | 35.1 (17.9)
  STAI - Trait Anxiety (range 20-80) Higher = more anxiety | 37.0 (11.5) | 34.8 (14.7)
  Maternal Confidence Questionnaire (range 0-56) Higher = more stress | 44.2 (9.0) | 49.1 (7.6)
  ICQ - Mom and Baby (range 0-5), Higher = better care | 4.3 (0.5) | 4.3 (0.8)
  ICQ - Emotionality (range 0-5), Higher = better care | 4.2 (0.9) | 4.3 (0.9)
  ICQ - Responsiveness (range 0-5), Higher = better care | 3.7 (0.8) | 4.1 (0.9)

8. Secondary Outcome: 1 Year Follow-Up Questionnaire
Description: The infant's mother completed a questionnaire with the following measures: the ASQ, SP-2, STAI, Beck Depression Inventory (BDI), PSI, Maternal Confidence Questionnaire (MCQ), ICQ, Pediatric Eating Assessment Tool (Pedi-eat), and Behavioral Pediatrics Feeding Assessment Scale (BPFAS). ASQ, SP-2, STAI, PSI, MCQ, and ICQ are previously described in discharge questionnaire outcome data. The BDI was used to measure maternal depression at time of follow-up. The Pedi-eat and BPFAS were used to assess infant feeding skills. Possible score ranges and directions of scores are reported below under each individual variable.
Time Frame: One year corrected age.
Population: Number of participants analyzed reflects the number of received follow-up questionnaires at 1 year corrected age. Participants who died, transferred to a different NICU prior to discharge, or did not complete follow-up questionnaires were not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 21 | 18
score on a scale
  PSI - Defensive Responding (range 7-35), Higher = more dysfunction | 11.9 (4.4) | 11.7 (7.0)
  PSI - Parental Distress (range 12-60), Higher = more dysfunction | 20.8 (7.8) | 20.6 (11.6)
  PSI - Difficult Child (range 12-60), higher = more dysfunction | 20.1 (6.3) | 17.8 (8.1)
  Beck Depression Inventory (range 0-63), Higher = more depression | 3.6 (4.1) | 3.9 (5.9)
  STAI - State Anxiety (range 20-80), Higher = more anxiety | 33.7 (9.6) | 28.9 (9.0)
  STAI - Trait Anxiety (range 20-80), Higher = more anxiety | 35.8 (9.3) | 28.8 (13.1)
  Maternal Confidence Questionnaire (range 0-56), Higher = more confidence | 51.4 (5.2) | 52.4 (3.2)
  ICQ - Mom and Baby (range 0-5), higher = better care | 4.2 (0.9) | 4.3 (0.9)
  ICQ - Emotionality (range 0-5), higher = better care | 4.1 (0.9) | 3.8 (1.7)
  ICQ - Responsiveness (range 0-5), higher = better care | 4.5 (1.0) | 4.6 (1.1)
  ASQ - Communication (range 0-60), Higher = better | 38.6 (18.1) | 48.6 (10.3)
  ASQ - Problem Solving (range 0-60), Higher = better | 35.8 (20.4) | 41.1 (14.2)
  ASQ - Gross Motor (range 0-60), Higher = better | 34.1 (22.6) | 42.8 (19.6)
  ASQ - Fine Motor (range 0-60), higher = better | 46.5 (10.4) | 47.8 (14.0)
  ASQ - Personal-Social (range 0-60), higher = better | 36.0 (17.8) | 40.3 (16.4)
  Sensory Profile - Touch (range 10-50), higher = more dysfunction | 16.9 (6.2) | 19.7 (4.3)
  Sensory Profile - Auditory (range 7-35), Higher = more dysfunction | 9.7 (4.6) | 9.7 (5.0)
  Sensory Profile - Visual (range 8-40), Higher = more dysfunction | 22.0 (4.3) | 21.6 (4.2)
  Sensory Profile - Movement Processing (range 6-30), Higher = more dysfunction | 18.8 (3.8) | 20.3 (2.9)
  Sensory Profile - Oral (range 7-35), higher = more dysfunction | 11.4 (4.7) | 10.6 (4.4)
  Sensory Profile - General (range 10-50), Higher = more dysfunction | 14.2 (6.6) | 13.9 (6.1)
  Sensory Profile - Behavior (range 6-30), Higher = more dysfunction | 10.6 (5.3) | 11.2 (3.6)
  Pediatric Eating Assessment Tool (range 0-390), Higher = more dysfunction | 54.1 (31.6) | 61.2 (28.7)
  Behavioral Pediatrics Feeding Assessment Scale (range 0-175), Higher = more dysfunction | 55.4 (16.2) | 51.0 (16.1)

9. Secondary Outcome: Mother-Infant Interaction (at 1 Year Follow-up)
Description: At one year follow-up, mother-infant interaction will be assessed through the interaction subscale of the Parental Stress Index (PSI). A score in this subscale can range from 12-60, with higher scores indicating a greater degree of dysfunction.
Time Frame: One year corrected age.
Population: Overall number of participants analyzed reflects the number of participants who returned completed questionnaires at 1 year corrected age. Reasons for lack of completion included: death of infant, transfer to different hospital prior to NICU discharge, lost to follow-up (not responding to calls/mail).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 21 | 18
score on a scale | 17.8 (6.2) | 14.3 (6.0)

10. Secondary Outcome: Parent Engagement During Hospitalization
Description: On each day of hospitalization (from birth to discharge, which often occurred close to term equivalent age; for an average of about 2 months), parents, health care professionals and the sensory support team documented the frequency of parent visitation, holding, and skin-to-skin care.
Time Frame: Every day of hospitalization (from birth through discharge, often close to term equivalent age; on average about 2 months).
Population: Overall number of participants analyzed reflects total number of participants with complete bedside logs at time of NICU discharge. Some participants were lost due to death or hospital transfer prior to discharge.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 28 | 24
Days
  Average number of days per 5-day week parents visited | 3.9 (1.3) | 3.9 (1.2)
  Average number of days per 5-day week parents held infant | 3.7 (1.1) | 3.7 (1.3)
  Average number of days per 5-day week parents provided skin-to-skin care | 1.6 (1.6) | 1.8 (1.7)

11. Secondary Outcome: Language Environmental Acquisition Device (LENA) Adult Word Count
Description: Audio recordings of a single 16 hour period to capture language and sound exposure occurred at 34 weeks using the Language Environmental Acquisition Device (LENA). The LENA device is a digital language processor that captures environmental sound for up to 16 hours and can quantify the number of adult words spoken during the 16 hour recording.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Control | Intervention
Number analyzed (Participants) | 17 | 12
words | 4618.1 (3934.0) | 4338.5 (4818.8)

12. Secondary Outcome: Percentage of Sensory Interventions Received
Description: Throughout hospitalization, parents, health care professionals and the sensory support team documented the type and amount of tactile and auditory exposures conducted. The percentage of recommended sensory doses that were received were documented.
Time Frame: Sensory exposures were documented every day of hospitalization (birth through discharge, often close to term) equivalent age).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of interventions received
Arm/Group | Control | Intervention
Number analyzed (Participants) | 28 | 24
percentage of interventions received | 80.5 (51.4) | 122.7 (34.9)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: No adverse events reported.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 3/39 | 1/31
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/31
Other Adverse Events (participants affected / at risk) | 0/39 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03316547/Prot_SAP_000.pdf